CLINICAL TRIAL: NCT01427842
Title: A Single-centred Randomised Trial of a New Vancomycin Dosing Method Compared to Standard Care in Everyday Patients Receiving Vancomycin
Brief Title: Dose Enhancement of Vancomycin IN Everyday Patients
Acronym: DEVINE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Canberra Hospital (Other)
Responsible Party: Principal Investigator, Kathryn Daveson, Dr Kathryn Daveson, The Canberra Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ETH.4.11.076
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Vancomycin Therapy
Keywords: Trough concentration; Vancomycin; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- DEVINE vancomycin regimen (Experimental): This is the intervention arm and will be the pharmacokinetically derived vancomycin dosing regimen.
  Interventions: Drug: DEVINE vancomycin regimen

INTERVENTIONS:
Drug: DEVINE vancomycin regimen — The dosing regimen varies by weight and height and by initial or ongoing dose prescribed. The loading dose is based on actual volume of distribution of vancomycin whilst the ongoing doses are based on creatinine clearance.
  Other Names: Pharmacokinetically derived vancomycin dosing regimen; Pharmacokinetic vancomycin regimen

SUMMARY:
Current Australian guidelines for vancomycin commonly underdoses individuals particularly in the first 48 hours.

The aim of the trial is to compare two dosing regimens; the current Australian guidelines versus a more appropriately modeled pharmacokinetic based regimen with the overall aim of developing a new vancomycin dosing strategy that will enable patients to have more individualised and therapeutically efficacious treatment.

The hypothesis is that dosing vancomycin according to a pharmacokinetically modeled regimen increases the likelihood of achieving therapeutic trough levels of vancomycin within the first 48 hours (or at steady state, whichever is sooner) compared to dosing vancomycin according to the current Antibiotic guidelines.

DETAILED DESCRIPTION:
DEVINE will be a randomised controlled trial of a new vancomycin dosing regimen against a control.

The control group regimen will receive the doses recommended by Therapeutic Guidelines - Antibiotics 2010. The intervention group will receive a dosing regimen that has been devised by modelling the antibiotic properties within the body over a large range of renal function and weight that will be more specific for the individual patient. They will receive this regimen for approximately 36-60 hours at which point they will have a vancomycin level blood test (a routine practice as part of their normal care). After this time the treating team will determine further dosing requirements.

All patients will be randomised at commencement of vancomycin with consent being obtained for the trial prior to the first dose of vancomycin

ELIGIBILITY:
Inclusion Criteria:

* All patients in general wards requiring routine treatment with vancomycin

Exclusion Criteria:

* GFR < 30mL/min(as measured by Cockcroft Gault equation)
* Age < 16 yrs
* Weight > 200kg
* Patients dosing with Vancomycin other than BD according to national guidelines (ie continuous infusions, q6h etc)
* Vancomycin infused at a rate other than 500mL/min

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Trough vancomycin concentration | At steady state for vancomycin received between 36 and 60 hours after the initial dose of vancomycin
  The primary outcome measure will be the trough serum vancomycin concentration measured at steady state usually between 36 and 60 hours after the initial dose of vancomycin. This according to Australian targets is between 12-18mg/L.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Daveson, Bsc, MBBS, MPH, Principal Investigator — The Canberra Hospital
Locations (1):
- The Canberra Hospital, Canberra, Australian Capital Territory, Australia